CLINICAL TRIAL: NCT02942745
Title: NIH-NCI U54 University of Guam/Cancer Center of Hawaii Partnership Full Project II: The Betel Nut Intervention Trial
Brief Title: Testing the Effectiveness of a Betel Nut Cessation Program
Acronym: BENIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guam (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Hawaii Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2U54CA143728 (NIH); 2U54CA143728 (NIH)
Record Dates: First submitted 2016-09-22; First posted 2016-10-24 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2019-11

CONDITIONS: Betel Nut Chewer; Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation

ARMS (2):
- Control (Placebo Comparator): Minimal interaction between participant and facilitator regarding cessation strategies. Participants will only be given a betel nut cessation booklet.
  Interventions: Behavioral: Betel Nut Cessation Booklet
- Experimental (Experimental): Intensive 5-session intervention program over the span of 22 days, with an additional follow up session after 6 months. The sessions will utilize betel nut cessation social support groups, as well as interactive discussion on how to quit chewing.
  Interventions: Behavioral: Betel Nut Cessation Social Support; Behavioral: Betel Nut Cessation Booklet

INTERVENTIONS:
Behavioral: Betel Nut Cessation Social Support — The cessation sessions will be led by trained facilitators over 22-day period. Session 1 (Day 1) includes a discussion of health risks associated with betel nut chewing, and introduction to self-monitoring and triggers logs. Session 2 (Day 8) includes a review of their logs, and discussions of lifestyle changes to assist cessation of betel nut chewing. Session 3 (Day 15) will be the quit day for chewers. Coping mechanisms and plans to maximize social support will be discussed. Session 4 (Day 18) will focus on quitting experiences. Facilitators will also review the negative health effects when wanting to chew again. Discussion on quitting experiences will continue in Session 5 (Day 22). Facilitators will also address those who have experienced relapse, and how to manage relapse.
  Arms: Experimental
Behavioral: Betel Nut Cessation Booklet — Participants will receive minimal intervention via a single booklet that contains all the information offered in the experimental group, minus the social support sessions. The participants will meet with study staff individually at a designated office in Guam or Saipan to receive the betel nut cessation booklet, complete three assessments (baseline, 22 days, 6 months), and provide saliva samples.

SUMMARY:
Areca nut, also known as betel nut, is the fourth most commonly consumed psychoactive substance in the world, following only alcohol, nicotine, and caffeine in prevalence of consumption. Although betel nut is chewed by approximately 600 million people globally, its use is concentrated in South Asia, Southeast Asia, and some Pacific Islands. Betel nut has been classified as a Group 1 carcinogen by the International Agency for Research on Cancer. Despite the global significance and carcinogenicity of betel nut, there has been very little behavioral or psychological research about betel nut chewing, and there has been no systematic research on the topic of betel nut cessation interventions. The current intervention builds directly upon the National Institutes of Health - National Cancer Institute's U54 University of Guam/University of Hawaii Cancer Center Comprehensive Partnership to Advance Health Equity. Previous data collected through the partnership suggest that betel nut chewers, like smokers, generally want and intend to quit, but do not have specific plans of how or when they will quit. In addition, most betel nut chewers in the partnership's previous study already have tried to quit on one or more occasions. The findings suggest that betel nut chewers could benefit from cessation programs modeled after smoking cessation programs. During 2014, partnership investigators conducted a feasibility study of the betel nut cessation program. The program was well received and yielded surprisingly high rates of self-reported betel nut cessation.

Specific Aim 1. To test the efficacy of an intensive group-based betel nut cessation program.

Specific Aim 2. To quantitatively determine the efficacy of the group-based betel nut cessation intervention trial using bio-verification.

DETAILED DESCRIPTION:
The general framework employed to guide the intervention is cognitive-behavioral therapy. The cognitive-behavioral therapy is goal-oriented and problem-focused. The goal of the intervention is to help betel nut chewers to quit chewing betel nut using structured sessions. The cognitive component addresses chewers' attitudes and beliefs about betel nut chewing. Preliminary data from a feasibility study revealed that most participants initially underestimated such negative health effects of betel nut. The behavioral component of the intervention aims to replace chewing-promoting behaviors with behaviors that are more conducive to quitting betel nut and staying quit, and preparing responses for social situations where pressure to chew is likely to occur.

The structure of the proposed betel nut cessation program is modeled after a specific group-based cognitive-behavioral smoking cessation program. The program was selected because it is a well-established and evidence-based group cessation program. The intervention will consist of a 22-day, five-session support and informational group program. Betel nut use will be evaluated via surveys and bio-verification at three points: at the initial group meeting, at the final group meeting, and six months following the final group meeting.

Group Intervention Format and Procedures

Five group sessions will be conducted over a period of 22 days per cohort. Group meetings will be approximately one hour in length and will be conducted by study investigators and staff. Surveys will be administered at the first and last group meetings, as well as six months after the last meeting. Surveys will be self-administered at the beginning of the intervention sessions. Confidentiality will be emphasized at all meetings, but especially so in the first session, and will be addressed specifically in the informed consent document. Participants will be reminded that participation is completely voluntary and that withdrawal without penalty is always an option. At most sessions, handouts will be provided and topical "homework" will be distributed.

Saliva Samples

Saliva samples (ca. 1-2 mL) for intervention condition participants will be collected at the same times as the three survey assessments (baseline, the final group intervention session, and the six-month follow-up). Saliva samples for control condition participants (also ca. 1-2 mL) will be collected on the same schedule as the intervention condition participants. From the saliva samples, Dr. Adrian Franke's laboratory will measure by liquid chromatography mass spectrometry levels of salivary biomarkers previously identified in the pilot study, which identified compounds specific for areca nuts and betel leaves that were extracted while chewing three different betel preparations. The studies also revealed that the compounds are secreted into saliva and appear in chewers' saliva up to eight hours after the chewing event. To verify self-reports of betel nut abstinence, the investigators will set cut-offs for levels of alkaloids specific for areca nuts as follows: arecoline 60 ng/mL, arecaidine 10 ng/mL, guvacoline 20 ng/mL, and guvacine 6 ng/mL). Levels above the values will indicate evidence of recent betel nut consumption. Participants whose saliva tests reveal values above the specified cut-offs will be considered current chewers for the purposes of bio-verified outcomes (i.e., chewer or non-chewer status). The biomarker results will be used to compare self-reports of recent chewing behavior (amount and recency) with biomarker data to assess dose-response effects.

Saliva samples will be collected in Guam and Saipan in 20 mL conical polypropylene tubes which will be initially stored at -20°C. Aggregated samples will be shipped to Hawaii via FedEx. Shipments will be performed whenever 50-60 samples are successfully collected. After arriving in Hawaii, samples will be stored in Dr. Adrian Franke's lab at -80°C until analysis. All samples available at Dr. Adrian Franke's lab will be analyzed in one batch at the end of each annual cycle of the study.

Survey Assessments

Baseline Survey

The baseline survey will be administered during the first group session. Saliva samples will be collected.

First Follow-Up Survey

The first follow-up survey will be administered during the final group session. Participants will indicate any attempt to quit chewing betel nut since starting the intervention program, current chewing status (chewer or ex-chewer), number of group sessions attended (and reasons for absence, if applicable), and quid composition (if still chewing). The participants will also be asked several questions to measure satisfaction with the cessation program. Saliva samples will be collected for a second time.

Second Follow-Up Survey

Six months post-cessation, participants will arrange to meet with study staff to complete a final survey assessment. Participants will be asked again to evaluate the program, as well as follow-up questions regarding current chewing status and betel quid composition. Saliva samples will be collected for a final time.

Measurement of Cessation Outcomes

Primary cessation outcomes will be assessed by self-reported 7-day point prevalence abstinence bio-verified by the saliva tests. Participants who self-report chewing cessation but who test positive for the betel nut biomarker will be classified as chewers.

Data Analysis

The data analysis plan was designed under the direct guidance of the U54 Biostatistics Core. The goal of the analysis is to determine if the proposed intervention strategy affects cessation of betel nut chewing. Information on chewing behavior will be collected at baseline, month 1, and month 6 for the intervention (IN0, IN1, IN6) and control conditions (C0, C1, C6). The efficacy of the cessation program will be assessed by estimation and comparison of cessation prevalence over time, defined as the proportion who are not chewing betel nut. The first test of efficacy will compare the cessation status between randomization groups at month 1 and month 6, using a logistic mixed model, which will account for the repeated (correlated) measures within each individual. The independent variables will include randomization group (defined as intent-to- treat), time (parameterized as two indicator variables), location (Guam/Saipan), and interaction terms between group and time. Potential confounders, such as gender, ethnicity and age, will be added to the models. The F-test for the interaction term for 6 months will be the test of efficacy. Statistics of interest from the model include the odds ratio and 95% confidence interval (CI) comparing randomization groups, and the covariate-adjusted probabilities of cessation and their 95% CIs, predicted by group from the model. The data will be analyzed within subgroups, such as location (Guam or Saipan) to provide information on whether the intervention was more effective in select groups. The investigators will model treatment as the number of sessions attended to determine if the program was more effective in more compliant participants. The mixed model uses all available data points at each time point. If there is evidence of non-random missingness, such as by differential drop-out between groups, multiple imputation will be used to determine if missing data led to biased results.

ELIGIBILITY:
Inclusion Criteria:

* Self-described betel nut chewer (chewed betel nut for at least 1 year, and at a rate of at least 3 days per week). Must chew a quid consisting of areca nut, slaked lime, betel leaf, tobacco, and/or other optional ingredients.
* Age ≥ 18 years
* Reside in Guam or Saipan
* Able to understand, speak, and read English
* Provide signed informed consent and agree to comply with all protocol-specified procedures (e.g., providing saliva samples, participating in five one-hour group sessions over a period of 22 days) and follow-up evaluations

Exclusion Criteria:

* Chews betel nut without tobacco
* Does not speak, read, and/or write English
* Women who are pregnant or nursing
* Psychiatric illness/social situations that would limit compliance with study requirements
* Other illness that in the opinion of the investigator would exclude the patient from participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in number of participants who self-report that they quit chewing betel nut to be measured via survey | 22 days
  This will measure cessation prevalence immediately after the program
Change in number of participants who self-report that they quit chewing betel nut to be measured via survey | 6 months
  This will measure cessation prevalence (stay-quit) long-term

SECONDARY OUTCOMES:
Levels of cotinine and betel nut biomarkers in saliva samples to be tested via liquid chromatography mass spectrometry | 22 days
  Cut-off levels for betel nut biomarkers include arecoline (60 ng/mL), arecaidine (10 ng/mL), guvacoline (20 ng/mL), and guvacine (6 ng/mL).
Levels of cotinine and betel nut biomarkers in saliva samples to be tested via liquid chromatography mass spectrometry | 6 months
  Cut-off levels for betel nut biomarkers include arecoline (60 ng/mL), arecaidine (10 ng/mL), guvacoline (20 ng/mL), and guvacine (6 ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Yvette C Paulino, PhD, CPH, Principal Investigator — University of Guam, University of Hawaii; Thaddeus A Herzog, PhD, Principal Investigator — University of Hawaii
Locations (1):
- University of Guam, Mangilao Village, Guam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benegal V, Rajkumar RP, Muralidharan K. Does areca nut use lead to dependence? Drug Alcohol Depend. 2008 Sep 1;97(1-2):114-21. doi: 10.1016/j.drugalcdep.2008.03.016. Epub 2008 May 19. PMID 18490113
- [Background] Chu NS. Neurological aspects of areca and betel chewing. Addict Biol. 2002 Jan;7(1):111-4. doi: 10.1080/13556210120091473. PMID 11900630
- [Background] Ghani WM, Razak IA, Yang YH, Talib NA, Ikeda N, Axell T, Gupta PC, Handa Y, Abdullah N, Zain RB. Factors affecting commencement and cessation of betel quid chewing behaviour in Malaysian adults. BMC Public Health. 2011 Feb 7;11:82. doi: 10.1186/1471-2458-11-82. PMID 21294919
- [Background] Gupta B, Johnson NW. Systematic review and meta-analysis of association of smokeless tobacco and of betel quid without tobacco with incidence of oral cancer in South Asia and the Pacific. PLoS One. 2014 Nov 20;9(11):e113385. doi: 10.1371/journal.pone.0113385. eCollection 2014. PMID 25411778
- [Background] Gupta PC, Ray CS. Epidemiology of betel quid usage. Ann Acad Med Singap. 2004 Jul;33(4 Suppl):31-6. PMID 15389304
- [Background] Gupta PC, Warnakulasuriya S. Global epidemiology of areca nut usage. Addict Biol. 2002 Jan;7(1):77-83. doi: 10.1080/13556210020091437. PMID 11900626
- [Background] Haddock RL. Oral cancer incidence disparity among ethnic groups on Guam. Pac Health Dialog. 2005 Mar;12(1):153-4. PMID 18181481
- [Background] Haddock RL, Whippy HJ, Talon RJ, Montano MV. Ethnic disparities in cancer incidence among residents of Guam. Asian Pac J Cancer Prev. 2009 Jan-Mar;10(1):57-62. PMID 19469625
- [Background] Herzog TA, Murphy KL, Little MA, Suguitan GS, Pokhrel P, Kawamoto CT. The Betel Quid Dependence Scale: replication and extension in a Guamanian sample. Drug Alcohol Depend. 2014 May 1;138:154-60. doi: 10.1016/j.drugalcdep.2014.02.022. Epub 2014 Feb 26. PMID 24629627
- [Background] IARC Working Group on the Evaluation of Carcinogenic Risks to Humans. Betel-quid and areca-nut chewing and some areca-nut derived nitrosamines. IARC Monogr Eval Carcinog Risks Hum. 2004;85:1-334. No abstract available. PMID 15635762
- [Background] IARC Working Group on the Evaluation of Carcinogenic Risks to Humans. Smokeless tobacco and some tobacco-specific N-nitrosamines. IARC Monogr Eval Carcinog Risks Hum. 2007;89:1-592. No abstract available. PMID 18335640
- [Background] Jeng JH, Chang MC, Hahn LJ. Role of areca nut in betel quid-associated chemical carcinogenesis: current awareness and future perspectives. Oral Oncol. 2001 Sep;37(6):477-92. doi: 10.1016/s1368-8375(01)00003-3. PMID 11435174
- [Background] Ko YC, Huang YL, Lee CH, Chen MJ, Lin LM, Tsai CC. Betel quid chewing, cigarette smoking and alcohol consumption related to oral cancer in Taiwan. J Oral Pathol Med. 1995 Nov;24(10):450-3. doi: 10.1111/j.1600-0714.1995.tb01132.x. PMID 8600280
- [Background] Lee CH, Ko YC, Huang HL, Chao YY, Tsai CC, Shieh TY, Lin LM. The precancer risk of betel quid chewing, tobacco use and alcohol consumption in oral leukoplakia and oral submucous fibrosis in southern Taiwan. Br J Cancer. 2003 Feb 10;88(3):366-72. doi: 10.1038/sj.bjc.6600727. PMID 12569378
- [Background] Little MA, Pokhrel P, Murphy KL, Kawamoto CT, Suguitan GS, Herzog TA. The reasons for betel-quid chewing scale: assessment of factor structure, reliability, and validity. BMC Oral Health. 2014 Jun 3;14:62. doi: 10.1186/1472-6831-14-62. PMID 24889863
- [Background] Murti PR, Bhonsle RB, Pindborg JJ, Daftary DK, Gupta PC, Mehta FS. Malignant transformation rate in oral submucous fibrosis over a 17-year period. Community Dent Oral Epidemiol. 1985 Dec;13(6):340-1. doi: 10.1111/j.1600-0528.1985.tb00468.x. PMID 3866655
- [Background] Nair U, Bartsch H, Nair J. Alert for an epidemic of oral cancer due to use of the betel quid substitutes gutkha and pan masala: a review of agents and causative mechanisms. Mutagenesis. 2004 Jul;19(4):251-62. doi: 10.1093/mutage/geh036. PMID 15215323
- [Background] Norton SA. Betel: consumption and consequences. J Am Acad Dermatol. 1998 Jan;38(1):81-8. doi: 10.1016/s0190-9622(98)70543-2. PMID 9448210
- [Background] Paulino YC, Novotny R, Miller MJ, Murphy SP. Areca (Betel) Nut Chewing Practices in Micronesian Populations. Hawaii J Public Health. 2011 Mar;3(1):19-29. PMID 25678943
- [Background] Pindborg JJ, Sirsat SM. Oral submucous fibrosis. Oral Surg Oral Med Oral Pathol. 1966 Dec;22(6):764-79. doi: 10.1016/0030-4220(66)90367-7. No abstract available. PMID 5224185
- [Background] Secretan B, Straif K, Baan R, Grosse Y, El Ghissassi F, Bouvard V, Benbrahim-Tallaa L, Guha N, Freeman C, Galichet L, Cogliano V; WHO International Agency for Research on Cancer Monograph Working Group. A review of human carcinogens--Part E: tobacco, areca nut, alcohol, coal smoke, and salted fish. Lancet Oncol. 2009 Nov;10(11):1033-4. doi: 10.1016/s1470-2045(09)70326-2. No abstract available. PMID 19891056
- [Background] Thomas S, Kearsley J. Betel quid and oral cancer: a review. Eur J Cancer B Oral Oncol. 1993 Oct;29B(4):251-5. doi: 10.1016/0964-1955(93)90044-f. No abstract available. PMID 11706417
- [Background] Wen CP, Tsai MK, Chung WS, Hsu HL, Chang YC, Chan HT, Chiang PH, Cheng TY, Tsai SP. Cancer risks from betel quid chewing beyond oral cancer: a multiple-site carcinogen when acting with smoking. Cancer Causes Control. 2010 Sep;21(9):1427-35. doi: 10.1007/s10552-010-9570-1. Epub 2010 May 11. PMID 20458529
- [Background] Brown, R. A. (2003). Intensive behavioral treatment. In D. B. Abrams (Ed.), The tobacco dependence treatment handbook : a guide to best practices (pp. 118-177). New York: Guilford Press.
- [Background] Little, R. J. A., & Rubin, D. B. (2002). Statistical analysis with missing data. New York: John Wiley & Sons.
- [Background] Uncangco, A. A., Badowski, G., David, A. M., Ehlert, M. B., Haddock, R. L., & Paulino, Y. C. (2012). First Guam BRFSS Report 2017-2010. Retrieved from Mangilao, GU:
- [Background] World Health Organization. (2012). Review of areca (betel) nut and tobacco use in the Pacific: a technical report. Geneva: World Health Organization.
- [Background] Boucher BJ, Mannan N. Metabolic effects of the consumption of Areca catechu. Addict Biol. 2002 Jan;7(1):103-10. doi: 10.1080/13556210120091464. PMID 11900629
- [Background] Lin CF, Wang JD, Chen PH, Chang SJ, Yang YH, Ko YC. Predictors of betel quid chewing behavior and cessation patterns in Taiwan aborigines. BMC Public Health. 2006 Nov 3;6:271. doi: 10.1186/1471-2458-6-271. PMID 17081309
- [Background] Oakley E, Demaine L, Warnakulasuriya S. Areca (betel) nut chewing habit among high-school children in the Commonwealth of the Northern Mariana Islands (Micronesia). Bull World Health Organ. 2005 Sep;83(9):656-60. Epub 2005 Sep 30. PMID 16211156
- [Background] Shah SM, Merchant AT, Luby SP, Chotani RA. Addicted schoolchildren: prevalence and characteristics of areca nut chewers among primary school children in Karachi, Pakistan. J Paediatr Child Health. 2002 Oct;38(5):507-10. doi: 10.1046/j.1440-1754.2002.00040.x. PMID 12354270
- [Background] Warnakulasuriya S. Areca nut use following migration and its consequences. Addict Biol. 2002 Jan;7(1):127-32. doi: 10.1080/13556210120091491. PMID 11900632
- [Background] Uncangco AA, Badowski G, David AM, Ehlert MB, Haddock RL, Paulino YC. First Guam BRFSS Report 2017-2010. Mangilao, GU: 2012
- [Background] Lee CH, Ko AM, Warnakulasuriya S, Ling TY, Sunarjo, Rajapakse PS, Zain RB, Ibrahim SO, Zhang SS, Wu HJ, Liu L, Kuntoro, Utomo B, Warusavithana SA, Razak IA, Abdullah N, Shrestha P, Shieh TY, Yen CF, Ko YC. Population burden of betel quid abuse and its relation to oral premalignant disorders in South, Southeast, and East Asia: an Asian Betel-quid Consortium Study. Am J Public Health. 2012 Mar;102(3):e17-24. doi: 10.2105/AJPH.2011.300521. Epub 2012 Jan 19. PMID 22390524
- [Background] 33. Fiore M, Jaen CR, Baker TB, Bailey WC, Benowitz NL, Curry SJ, Dorfman SF, Froelicher ES, Goldstein MG, Healton CG, Henderson PN, Heyman RB, Koh HK, Kottke TE, Lando HA, Mecklenburg RE, Mermelstein RJ, Mullen PD, Orleans CT, Robinson L, Stitzer ML, Tommasello AC, Villejo L, Wewers ME. Treating Tobacco Use and Dependence: 2008 Update. Clinical Practice Guideline. 2008 update ed. Rockville, Md.: U.S. Dept. of Health and Human Services, Public Health Service; 2008. xvii, 256 p. p.
- [Background] Herzog TA. Analyzing the transtheoretical model using the framework of Weinstein, Rothman, and Sutton (1998): the example of smoking cessation. Health Psychol. 2008 Sep;27(5):548-56. doi: 10.1037/0278-6133.27.5.548. PMID 18823181
- [Background] Herzog TA, Pokhrel P. Ethnic differences in smoking rate, nicotine dependence, and cessation-related variables among adult smokers in Hawaii. J Community Health. 2012 Dec;37(6):1226-33. doi: 10.1007/s10900-012-9558-8. PMID 22438074
- [Background] Glover E, Wang M, WGlover P. Development of a high school smokeless tobacco cessation manual. Health Values: The Journal of Health Behavior, Education & Promotion. 1994;18(2):1-7.
- [Background] Williams S, Arheart KL, WKiesges R. A smokeless tobacco cessation program for postsecondary students. Health Values: The Journal of Health Behavior, Education & Promotion. 1995;19(3):1-9.
- [Background] Paulino Y. Betel nut chewing in Micronesian populations. Achievement Rewards for College Scientists Selection Meeting; 2008; Honolulu, HI.
- [Background] Paulino YC, Hurwitz EL. Making the case for clearly defining tobacco use in areca (betel) nut chewers. American Public Health Association Annual Meeting; 2014; New Orleans, LA
- [Background] Paulino YC, Hurwitz EL, Warnakulasuriya S, Gatewood RR, Pierson KD, Tenorio LF, Novotny R, Palafox NA, Wilkens LR, Badowski G. Screening for oral potentially malignant disorders among areca (betel) nut chewers in Guam and Saipan. BMC Oral Health. 2014 Dec 11;14:151. doi: 10.1186/1472-6831-14-151. PMID 25495475
- [Background] Paulino YC, Hurwitz EL, Wilkens LR, Novotny R, Miller MJ, Quinata KM. Pattern of areca (betel) nut chewing and obesity measures in Guam and Saipan, Mariana Islands. 20th International Epidemiologic Association World Congress of Epidemiology; 2014; Anchorage, AK.
- [Background] Chandra PS, Carey MP, Carey KB, Jairam KR. Prevalence and correlates of areca nut use among psychiatric patients in India. Drug Alcohol Depend. 2003 Apr 1;69(3):311-6. doi: 10.1016/s0376-8716(02)00329-0. PMID 12633917
- [Background] Mubeen K, Kumar CN, Puja R, Jigna VR, Chandrashekar H. Psychiatric morbidity among patients with oral sub-mucous fibrosis: a preliminary study. J Oral Pathol Med. 2010 Nov;39(10):761-4. doi: 10.1111/j.1600-0714.2010.00948.x. Epub 2010 Oct 4. PMID 20923447
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders : DSM-IV-TR. 4th ed. Washington, DC: American Psychiatric Association; 2000. xxxvii, 943 p. p.
- [Background] World Health Organization. The ICD-10 classification of mental and behavioural disorders : clinical descriptions and diagnostic guidelines. Geneva: World Health Organization; 1992. xii, 362 p. p.
- [Background] Winstock A. Areca nut-abuse liability, dependence and public health. Addict Biol. 2002 Jan;7(1):133-8. doi: 10.1080/13556210120091509. PMID 11900633
- [Background] Bhat SJ, Blank MD, Balster RL, Nichter M, Nichter M. Areca nut dependence among chewers in a South Indian community who do not also use tobacco. Addiction. 2010 Jul;105(7):1303-10. doi: 10.1111/j.1360-0443.2010.02952.x. PMID 20642513
- [Background] Lee CY, Chang CS, Shieh TY, Chang YY. Development and validation of a self-rating scale for betel quid chewers based on a male-prisoner population in Taiwan: the Betel Quid Dependence Scale. Drug Alcohol Depend. 2012 Feb 1;121(1-2):18-22. doi: 10.1016/j.drugalcdep.2011.07.027. Epub 2011 Sep 28. PMID 21955360
- [Background] Berlin I, Singleton EG, Pedarriosse AM, Lancrenon S, Rames A, Aubin HJ, Niaura R. The Modified Reasons for Smoking Scale: factorial structure, gender effects and relationship with nicotine dependence and smoking cessation in French smokers. Addiction. 2003 Nov;98(11):1575-83. doi: 10.1046/j.1360-0443.2003.00523.x. PMID 14616184
- [Background] Brandon TH, Baker TB. The Smoking Consequences Questionnaire: the subjective expected utility of smoking in college students. Psychological Assessment. 1991;3:484-91.
- [Background] Piper ME, Piasecki TM, Federman EB, Bolt DM, Smith SS, Fiore MC, Baker TB. A multiple motives approach to tobacco dependence: the Wisconsin Inventory of Smoking Dependence Motives (WISDM-68). J Consult Clin Psychol. 2004 Apr;72(2):139-54. doi: 10.1037/0022-006X.72.2.139. PMID 15065950
- [Background] Little MA, Pokhrel P, Murphy KL, Kawamoto CT, Suguitan GS, Herzog TA. Intention to quit betel quid: a comparison of betel quid chewers and cigarette smokers. Oral Health Dent Manag. 2014 Jun;13(2):512-8. PMID 24984674
- [Background] Franke AA, Morimoto Y, Yeh LM, Maskarinec G. Urinary isoflavonoids as a dietary compliance measure among premenopausal women. Asia Pac J Clin Nutr. 2006;15(1):88-94. PMID 16500883
- [Background] Le Marchand L, Hankin JH, Carter FS, Essling C, Luffey D, Franke AA, Wilkens LR, Cooney RV, Kolonel LN. A pilot study on the use of plasma carotenoids and ascorbic acid as markers of compliance to a high fruit and vegetable dietary intervention. Cancer Epidemiol Biomarkers Prev. 1994 Apr-May;3(3):245-51. PMID 8019375
- [Background] Franke AA, Mendez AJ, Lai JF, Arat-Cabading C, Li X, Custer LJ. Composition of betel specific chemicals in saliva during betel chewing for the identification of biomarkers. Food Chem Toxicol. 2015 Jun;80:241-246. doi: 10.1016/j.fct.2015.03.012. Epub 2015 Mar 19. PMID 25797484
- [Background] Franke AA, Lai JF, Kawamoto CT, Pokhrel P, Herzog TA. University of Hawai'i Cancer Center connection: Areca (betel) nut consumption: an underappreciated cause of cancer. Hawaii J Med Public Health. 2014 Dec;73(12):400-3. No abstract available. PMID 25628974
- [Background] Friedman LM, Furberg C, DeMets DL. Fundamentals of clinical trials. 3rd ed. New York: Springer; 1998. xviii, 361 p. p.
- [Background] Borrelli B. The assessment, monitoring, and enhancement of treatment fidelity in public health clinical trials. J Public Health Dent. 2011 Winter;71 Suppl 1:S52-63. PMID 21656954
- [Background] Perkins KA, Conklin CA, Levine MD. Cognitive-behavioral therapy for smoking cessation : a practical guidebook to the most effective treatments. New York: Routledge; 2008. xxii, 258 p. p.
- [Background] Brown RA. Intensive behavioral treatment. In: Abrams DB, editor. The tobacco dependence treatment handbook : a guide to best practices. New York: Guilford Press; 2003. p. 118-77.
- [Background] Stead LF, Lancaster T. Group behaviour therapy programmes for smoking cessation. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001007. doi: 10.1002/14651858.CD001007.pub2. PMID 15846610
- [Background] Little RJA, Rubin DB. Statistical analysis with missing data. New York: John Wiley & Sons; 2002.
- [Background] Cohen J. Statistical power analysis for the behavioral sciences. 2nd ed. Hillsdale, N.J.: L. Erlbaum Associates; 1988. xxi, 567 p. p.
- [Background] Lord GA, Lim CK, Warnakulasuriya S, Peters TJ. Chemical and analytical aspects of areca nut. Addict Biol. 2002 Jan;7(1):99-102. doi: 10.1080/13556210120091455. PMID 11900628
- [Result] Boyle RG, Enstad C, Asche SE, Thoele MJ, Sherwood NE, Severson HH, Ebbert J, Solberg LI. A randomized controlled trial of Telephone Counseling with smokeless tobacco users: the ChewFree Minnesota study. Nicotine Tob Res. 2008 Sep;10(9):1433-40. doi: 10.1080/14622200802279872. PMID 19023834
- [Result] Walsh MM, Langer TJ, Kavanagh N, Mansell C, MacDougal W, Kavanagh C, Gansky SA. Smokeless tobacco cessation cluster randomized trial with rural high school males: intervention interaction with baseline smoking. Nicotine Tob Res. 2010 Jun;12(6):543-50. doi: 10.1093/ntr/ntq022. Epub 2010 May 3. PMID 20439384
- [Derived] Rojas GA, Erari S, Paulino YC, Herzog TA. Facilitator experiences and lessons learned from the Betel nut intervention trial (BENIT). BMC Public Health. 2024 Jan 24;24(1):288. doi: 10.1186/s12889-024-17788-4. PMID 38267890
- [Derived] Herzog TA, Wilkens LR, Badowski G, Mendez AJP, Franke AA, Pokhrel P, Chennaux JSN, Tenorio LF, Sotto PP, Kawamoto CT, Paulino YC. The Betel Nut Intervention Trial (BENIT)-A Randomized Clinical Trial for Areca Nut and Betel Quid Cessation: Primary Outcomes. Int J Environ Res Public Health. 2023 Aug 21;20(16):6622. doi: 10.3390/ijerph20166622. PMID 37623205